CLINICAL TRIAL: NCT00399035
Title: A Randomised, Double-blind, Phase III Study to Compare the Efficacy and Safety of Cediranib (AZD2171, RECENTIN™) When Added to 5 Fluorouracil, Leucovorin and Oxaliplatin (FOLFOX) or Capecitabine and Oxaliplatin (XELOX) With the Efficacy and Safety of Placebo When Added to FOLFOX or XELOX in Patients With Previously Untreated Metastatic Colorectal Cancer.
Brief Title: Cediranib (AZD2171, RECENTIN™) in Addition to Chemotherapy in Patients With Untreated Metastatic Colorectal Cancer
Acronym: HORIZON II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00051; EUDRACT No 2006-001194-14; HORIZON II
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Cediranib; RECENTIN
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cediranib; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Infusions, Intravenous; XELOX; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- FOLFOX + placebo Cediranib (Placebo Comparator): FOLFOX + placebo Cediranib
  Interventions: Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin); Drug: Cediranib Placebo
- Xelox + placebo Cediranib (Placebo Comparator): Xelox + placebo Cediranib
  Interventions: Drug: XELOX (Capecitabine and Oxaliplatin); Drug: Cediranib Placebo
- FOLFOX + Cediranib (Experimental): FOLFOX + Cediranib
  Interventions: Drug: Cediranib; Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin)
- XELOX + Cediranib (Experimental): XELOX + Cediranib
  Interventions: Drug: Cediranib; Drug: XELOX (Capecitabine and Oxaliplatin)

INTERVENTIONS:
Drug: Cediranib — oral tablet
  Other Names: AZD2171; RECENTIN™
  Arms: FOLFOX + Cediranib; XELOX + Cediranib
Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin) — intravenous infusion
  Other Names: Other Names:; 5-FU; Drug: Leucovorin (in FOLFOX); intravenous infusion; Drug: Oxaliplatin (in FOLFOX); Eloxatin®
  Arms: FOLFOX + Cediranib; FOLFOX + placebo Cediranib
Drug: XELOX (Capecitabine and Oxaliplatin) — intravenous oxaliplatin 130 mg/ m^2(day 1) followed by oral capecitabine 1,000 mg/ m^2twice daily (day 1 to day 15)
  Other Names: Xeloda® + Eloxatin®
  Arms: XELOX + Cediranib; Xelox + placebo Cediranib
Drug: Cediranib Placebo — oral tablet
  Arms: FOLFOX + placebo Cediranib; Xelox + placebo Cediranib

SUMMARY:
The purpose of this study is to determine if Cediranib when added to chemotherapy is more effective than chemotherapy alone in prolonging life expectancy and slowing disease progression in patients with previously untreated metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Carcinoma of the colon or rectum
* One or more measurable lesions

Exclusion Criteria:

* Adjuvant/neoadjuvant therapy within 6-12 months of study entry
* Untreated unstable brain or meningeal metastases
* Specific laboratory ranges
* Specific cardiovascular problems
* Participation in other trials within 30 days

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca
Locations (90):
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Resistencia
  - Research Site, Rosario
  - Research Site, Santa Fe
- Australia (7):
  - Research Site, Ashford
  - Research Site, Camperdown
  - Research Site, Heidelberg
  - Research Site, Hornsby
  - Research Site, Liverpool
  - Research Site, Waratah
  - Research Site, Wodonga
- Brazil (8):
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
- Bulgaria (6):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- China (11):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Tianjin
- Czechia (12):
  - Research Site, Brno
  - Research Site, Cheb
  - Research Site, České Budějovice
  - Research Site, Jičín
  - Research Site, Jihlava
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Pribram - Zdabor
  - Research Site, Šumperk
  - Research Site, Zlín
  - Research Site, Znojmo
- Germany (6):
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Goslar
  - Research Site, Hamburg
  - Research Site, Hildesheim
  - Research Site, Mannheim
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Szombathely
  - Research Site, Zalaegerszeg
- India (2):
  - Research Site, Hyderabad
  - Research Site, Trivandrum
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Quezon
  - Research Site, Quezon City
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Torun
  - Research Site, Wroclaw
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Switzerland (4):
  - Research Site, Bellinzona
  - Research Site, Lausanne
  - Research Site, Locarno
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (4):
  - Research Site, Aberdeen
  - Research Site, Belfast
  - Research Site, Leicester
  - Research Site, Manchester

REFERENCES:
- [Derived] Smith JC, Brooks L, Hoff PM, McWalter G, Dearden S, Morgan SR, Wilson D, Robertson JD, Jurgensmeier JM. KRAS mutations are associated with inferior clinical outcome in patients with metastatic colorectal cancer, but are not predictive for benefit with cediranib. Eur J Cancer. 2013 Jul;49(10):2424-32. doi: 10.1016/j.ejca.2013.02.023. Epub 2013 Mar 16. PMID 23510802
- See also: CSR-D8480C00051.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=424&filename=CSR-D8480C00051.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised=full analysis set: Cediranib 20mg=502, Placebo=358; Safety set: Cediranib 20mg=500, Cediranib 30mg=214, Placebo=358
Pre-assignment Details: Cediranib 30 mg discontinued following Phase II, Cediranib 20 mg chosen dose for comparing with Placebo.
  1254 patients enrolled to the study, 1076 recieved study treatment; 2 patients lost for Cediranib 20 mg/day, and 2 patients lost for Cediranib 30 mg/day.The 4 patients that didn't receive drug are intentionally included.
Groups:
- Cediranib 20 mg/Day: [Cediranib 20mg/day+FOLFOX/XELOX].2 FOLFOX regimens were chosen:FOLFOX4 or mFOLFOX6(repeated every 2 weeks.FOLFOX4:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 200mg/m2(or equivalent folinic acid preparation) by iv infusion over 2h on Day1 and Day2;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1 and Day2;5-FU 600 mg/m2 immediately after the 5-FU bolus dosed by continuous iv infusion over 22h on Day1 and Day2.mFOLFOX6:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 400mg/m2(or equivalent folinic acid preparation)dosed iv over 2h on Day1;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1,followed immediately by 5-FU 2400mg/m2 dosed by continuous iv infusion over 46h.XELOX:The XELOX regimen was to be repeated every 3 weeks:oxaliplatin 130mg/m2 dosed by iv infusion over 2h on Day1;capecitabine 1000mg/m2 orally twice daily on Days1 to 14.
- Cediranib 30 mg/Day: [Cediranib 30mg/day+FOLFOX/XELOX].2 FOLFOX regimens were chosen:FOLFOX4 or mFOLFOX6(repeated every 2 weeks.FOLFOX4:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 200mg/m2(or equivalent folinic acid preparation) by iv infusion over 2h on Day1 and Day2;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1 and Day2;5-FU 600 mg/m2 immediately after the 5-FU bolus dosed by continuous iv infusion over 22h on Day1 and Day2.mFOLFOX6:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 400mg/m2(or equivalent folinic acid preparation)dosed iv over 2h on Day1;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1,followed immediately by 5-FU 2400mg/m2 dosed by continuous iv infusion over 46h.XELOX:The XELOX regimen was to be repeated every 3 weeks:oxaliplatin 130mg/m2 dosed by iv infusion over 2h on Day1;capecitabine 1000mg/m2 orally twice daily on Days1 to 14.
- Placebo: [Placebo +FOLFOX/XELOX].2 FOLFOX regimens were chosen:FOLFOX4 or mFOLFOX6(repeated every 2 weeks.FOLFOX4:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 200mg/m2(or equivalent folinic acid preparation) by iv infusion over 2h on Day1 and Day2;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1 and Day2;5-FU 600 mg/m2 immediately after the 5-FU bolus dosed by continuous iv infusion over 22h on Day1 and Day2.mFOLFOX6:oxaliplatin 85mg/m2 dosed by iv infusion over 2h on Day1;leucovorin 400mg/m2(or equivalent folinic acid preparation)dosed iv over 2h on Day1;5-FU 400mg/m2 iv bolus immediately after completion of the oxaliplatin/leucovorin infusion on Day1,followed immediately by 5-FU 2400mg/m2 dosed by continuous iv infusion over 46h.XELOX:The XELOX regimen was to be repeated every 3 weeks:oxaliplatin 130mg/m2 dosed by iv infusion over 2h on Day1;capecitabine 1000mg/m2 orally twice daily on Days1 to 14.
Period: Overall Study
Arm/Group | Cediranib 20 mg/Day | Cediranib 30 mg/Day | Placebo
Started | 502 | 216 | 358
Completed | 189 | 58 | 106
Not Completed | 313 | 158 | 252
Not completed — Death | 289 | 141 | 234
Not completed — Lost to Follow-up | 2 | 1 | 5
Not completed — Withdrawal by Subject | 19 | 15 | 12
Not completed — Incorrect enrolment/eligib not fulfilled | 1 | 0 | 1
Not completed — Severe non-compliance with protocol | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cediranib 20 mg: Cediranib 20 mg + FOLFOX/XELOX
- Placebo: Placebo + FOLFOX/XELOX
- Cediranib 30 mg: Cediranib 30 mg/day + FOLFOX/XELOX
- Total: Total of all reporting groups
Arm/Group | Cediranib 20 mg | Placebo | Cediranib 30 mg | Total
Number analyzed (Participants) | 502 | 358 | 216 | 1076
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 57.8 (11.14) | 57.2 (11.63) | 59.4 (10.69) | 57.6 (11.34)
Gender [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 203 | 146 | 93 | 442
    Male | 299 | 212 | 123 | 634

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: RECIST criteria defined as follows: Target lesions Complete Response (CR) Disappearance of all target lesions Partial Response (PR) At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD.Progressive Disease (PD) At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded (either at baseline or at previous assessment since treatment began).Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Non-target lesions Complete Response (CR) Disappearance of all non-target lesions Non-Complete Response (non-CR/Non- Progression [non-PD]) Persistence of one or more non-target lesion or/and maintenance of tumour marker level above the normal limits. Progression (PD) Unequivocal progression of existing nontarget lesions.
Time Frame: RECIST assessed at baseline every 6 weeks through to week 24 and 12 week thereafter through to progression or data cut off date of 21/03/10 whichever was earliest.
Population: Two cediranib doses (20 mg and 30 mg) were initially included in this study; however, it was intended that one dose would be selected for continuation.The decision was taken to continue with cediranib 20 mg. All efficacy analyses compared cediranib 20mg to placebo. No statistical analyses were performed on the 30mg group.
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Cediranib 20 mg: Cediranib 20 mg/day + FOLFOX/XELOX
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 502 | 358
Months | 8.6 [5.5 to 12.1] | 8.2 [4.1 to 11.1]

2. Primary Outcome: Overall Survival
Description: Number of months from randomisation to the date of death from any cause
Time Frame: Baseline through to date of death upto and including data cut off date of 21/03/10
Population: Two cediranib doses (20 mg and 30 mg) were initially included in this study; however, it was intended that one dose would be selected for continuation. The decision was taken to continue with cediranib 20 mg. All efficacy analyses compared cediranib 20mg to placebo. No statistical analyses were performed on the 30mg group.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 502 | 358
Months | 19.7 [11.0 to 36.1] | 18.9 [11.0 to 28.9]

3. Secondary Outcome: Overall Response Rate
Description: Objective tumour response(defined as a confirmed response of CR or PR).The definition for a confirmed response was met when an initial RECIST response of PR/CR was confirmed at the next scheduled visit as a PR/CR according to an evaluable assessment.Intervening assessments of non-evaluable or stable disease were allowable as long as the initial RECIST response was confirmed.RECIST criteria defined as follows: Target lesions Complete Response(CR)Disappearance of all target lesions Partial Response (PR).At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD. Progressive Disease (PD) At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded (either at baseline or at previous assessment since treatment began).Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.Non-target lesions Complete Response (CR) Disappearance of all non-target lesi
Time Frame: Baseline through to date of death upto and including data cut off date of 21/03/10
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 502 | 358
Participants | 254 | 178

4. Secondary Outcome: Best Percentage Change in Tumour Size
Description: Maximum percentage reduction or minimum percentage increase in tumour size where size is the sum of the longest diameters of the target lesions
Time Frame: Baseline through to date of death upto and including data cut off date of 21/03/10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage [change in tumour size (mm) ]
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 474 | 339
Percentage [change in tumour size (mm) ] | -42.49 (28.139) | -40.61 (31.992)

5. Secondary Outcome: Duration of Response
Description: Based on RECIST measurements taken throughout the study and best objective tumour response at the defined analysis cut-off point. Measured from the time the criteria for CR/PR are first met (whichever is recorded first) until the patient progresses or dies.
Time Frame: Treatment period from initial response up until data cut-off date of 21/03/10
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 254 | 178
Months | 8.5 [5.9 to 12.7] | 6.9 [4.8 to 11.0]

6. Secondary Outcome: Rate of Resection of Liver Metastases
Description: Number of patients undergoing liver resection, based on patients with liver disease at baseline
Time Frame: Post-randomisation until end of study
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 387 | 271
Participants | 21 | 17

7. Secondary Outcome: Time to Wound Healing Complications
Description: Number of days from post-randomisation surgery until wound healing complications
Time Frame: Post-randomisation until end of study
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Cediranib 20 mg | Placebo
Number analyzed (Participants) | 94 | 79
Days | 18 [1 to 93] | 18 [0 to 114]

ADVERSE EVENTS:
Groups:
- Cediranib 30mg: Cediranib 30mg/day + Folfox/Xelox
- Cediranib 20mg: Cediranib 20mg/day + Folfox/Xelox
Arm/Group | Cediranib 30mg | Cediranib 20mg | Placebo
Serious Adverse Events (participants affected / at risk) | 94/214 | 204/500 | 105/358
Other Adverse Events (participants affected / at risk) | 209/214 | 485/500 | 341/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30mg (N=214) | Cediranib 20mg (N=500) | Placebo (N=358)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 11 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Coombs Positive Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 2 | 3
Myocardial Infarction (Cardiac disorders) | 3 | 1 | 0
Cardiac Failure (Cardiac disorders) | 2 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 2 | 1
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 34 | 11
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 8 | 4
Vomiting (Gastrointestinal disorders) | 5 | 7 | 8
Ileus (Gastrointestinal disorders) | 1 | 5 | 4
Constipation (Gastrointestinal disorders) | 0 | 4 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 1
Subileus (Gastrointestinal disorders) | 3 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Fistula (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Fistula (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mechanical Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Proctocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 5 | 4
Asthenia (General disorders) | 1 | 1 | 3
Fatigue (General disorders) | 2 | 3 | 0
Death (General disorders) | 2 | 1 | 1
General Physical Health Deterioration (General disorders) | 1 | 1 | 0
Infusion Site Irritation (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 1
Performance Status Decreased (General disorders) | 1 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 2 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1 | 1
Hepatorenal Failure (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 3
Drug Hypersensitivity (Immune system disorders) | 1 | 3 | 2
Hypersensitivity (Immune system disorders) | 1 | 2 | 0
Food Allergy (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 7 | 8
Urinary Tract Infection (Infections and infestations) | 0 | 6 | 2
Sepsis (Infections and infestations) | 3 | 4 | 3
Gastroenteritis (Infections and infestations) | 2 | 3 | 0
Septic Shock (Infections and infestations) | 0 | 3 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 1
Abdominal Wall Abscess (Infections and infestations) | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0
Amoebic Dysentery (Infections and infestations) | 1 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0
Blastocystis Infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Campylobacter Intestinal Infection (Infections and infestations) | 0 | 1 | 0
Catheter Related Infection (Infections and infestations) | 1 | 1 | 1
Catheter Sepsis (Infections and infestations) | 0 | 1 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0 | 0
Central Line Infection (Infections and infestations) | 0 | 1 | 1
Colostomy Infection (Infections and infestations) | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1 | 0
Infected Epidermal Cyst (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Lung Abscess (Infections and infestations) | 1 | 0 | 0
Meningitis Bacterial (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1 | 0
Scrotal Abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 2 | 4
Comminuted Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Peroneal Nerve Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stent Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bilirubin Conjugated Increased (Investigations) | 0 | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 14 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign Neoplasm Of Spinal Cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Penis Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 4 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 3 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0
Central Nervous System Lesion (Nervous system disorders) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Nervous System Disorder (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neurological Symptom (Nervous system disorders) | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 1
Confusional State (Psychiatric disorders) | 1 | 1 | 1
Personality Change Due To A General Medical Condition (Psychiatric disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 5 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 3 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 3 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 2 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1 | 1
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 3 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysaesthesia Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 8 | 6 | 2
Deep Vein Thrombosis (Vascular disorders) | 2 | 3 | 1
Aortic Thrombosis (Vascular disorders) | 1 | 0 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral Embolism (Vascular disorders) | 0 | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30mg (N=214) | Cediranib 20mg (N=500) | Placebo (N=358)
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 139 | 84
Neutropenia (Blood and lymphatic system disorders) | 49 | 138 | 75
Leukopenia (Blood and lymphatic system disorders) | 15 | 84 | 39
Anaemia (Blood and lymphatic system disorders) | 24 | 40 | 43
Granulocytopenia (Blood and lymphatic system disorders) | 3 | 28 | 9
Hypothyroidism (Endocrine disorders) | 28 | 42 | 8
Diarrhoea (Gastrointestinal disorders) | 147 | 346 | 165
Nausea (Gastrointestinal disorders) | 92 | 256 | 169
Vomiting (Gastrointestinal disorders) | 83 | 230 | 126
Abdominal Pain (Gastrointestinal disorders) | 32 | 134 | 78
Stomatitis (Gastrointestinal disorders) | 59 | 118 | 48
Constipation (Gastrointestinal disorders) | 34 | 85 | 78
Abdominal Pain Upper (Gastrointestinal disorders) | 24 | 58 | 28
Dyspepsia (Gastrointestinal disorders) | 18 | 35 | 20
Abdominal Distension (Gastrointestinal disorders) | 6 | 27 | 19
Flatulence (Gastrointestinal disorders) | 4 | 27 | 12
Fatigue (General disorders) | 80 | 200 | 104
Pyrexia (General disorders) | 31 | 76 | 60
Asthenia (General disorders) | 32 | 74 | 45
Oedema Peripheral (General disorders) | 22 | 53 | 46
Drug Hypersensitivity (Immune system disorders) | 6 | 24 | 19
Urinary Tract Infection (Infections and infestations) | 15 | 40 | 14
Weight Decreased (Investigations) | 28 | 63 | 18
Alanine Aminotransferase Increased (Investigations) | 11 | 33 | 15
Aspartate Aminotransferase Increased (Investigations) | 9 | 33 | 18
Platelet Count Decreased (Investigations) | 6 | 33 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 92 | 229 | 125
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 58 | 22
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 14 | 48 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 17 | 41 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 34 | 14
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 22 | 12
Peripheral Sensory Neuropathy (Nervous system disorders) | 45 | 141 | 89
Paraesthesia (Nervous system disorders) | 49 | 97 | 85
Neuropathy Peripheral (Nervous system disorders) | 24 | 77 | 64
Headache (Nervous system disorders) | 35 | 70 | 34
Dizziness (Nervous system disorders) | 19 | 52 | 23
Hypoaesthesia (Nervous system disorders) | 7 | 38 | 17
Dysgeusia (Nervous system disorders) | 14 | 26 | 25
Dysaesthesia (Nervous system disorders) | 13 | 16 | 11
Insomnia (Psychiatric disorders) | 15 | 50 | 27
Proteinuria (Renal and urinary disorders) | 20 | 60 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 39 | 67 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 | 63 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 50 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 29 | 24
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 28 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 23 | 8
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 53 | 123 | 57
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 38 | 22
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 | 34 | 25
Rash (Skin and subcutaneous tissue disorders) | 9 | 33 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 14 | 16 | 11
Hypertension (Vascular disorders) | 96 | 226 | 41
Phlebitis (Vascular disorders) | 7 | 19 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.